CLINICAL TRIAL: NCT07227480
Title: Advancing Lung Cancer Screening One Text at a Time
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Francisco Cartujano, MD, Assistant Professor - Department of Public Health Sciences (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: STUDY00010975
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer Screening
Keywords: Lung Cancer Screening

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UR Screened (Experimental): A text messaging program designed to promote lung cancer screening
  Interventions: Behavioral: Text messaging program
- Control group (Active Comparator): A mailed educational material along with a flyer for the lung cancer screening program
  Interventions: Behavioral: Educational material

INTERVENTIONS:
Behavioral: Text messaging program — A text messaging program designed to promote lung cancer screening
  Arms: UR Screened
Behavioral: Educational material — A mailed educational material along with a flyer for the lung cancer screening program
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the feasibility, acceptability, and preliminary impact of text messaging to promote lung cancer screening.

DETAILED DESCRIPTION:
We will conduct a two-arm pilot randomized controlled trial with 40 adults. Participants will be randomized in a 1:1 ratio to either UR Screened (a text messaging program designed to promote lung cancer screening) or a control group (a mailed educational material along with a flyer for the lung cancer screening program). We will assess recruitment and follow-up rates, satisfaction with the program or educational material, and uptake of lung cancer screening at week 12. Additionally, we will compare screening rates between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 80 years old
* have not completed their annual screening for lung cancer
* have a 20 pack-year smoking history
* currently smoke or have quit within the past 15 years
* speak English and/or Spanish
* have a functioning cellphone number with unlimited text messaging capacity
* be willing to complete a baseline and a follow-up (at Month 3) survey

Exclusion Criteria:

* being up-to-date on their annual lung cancer screening

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants Who Undergo Lung Cancer Screening | Month 3
  The proportion of study participants who complete a lung cancer screening test within 3 months of study enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States